CLINICAL TRIAL: NCT02740179
Title: Mineralocorticoid Receptor Antagonism for Cardiovascular Health in HIV--The MIRACLE HIV Study
Brief Title: Effects of Eplerenone on Cardiovascular Disease in HIV (MIRACLE HIV Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P000464
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: HIV
Keywords: Eplerenone; Cardiovascular Disease; Mineralocorticoid Receptor Antagonist; Coronary Vasculature; Myocardial Inflammation; Myocardial Fibrosis; Atherosclerosis; Aldosterone
MeSH Terms: conditions — Cardiovascular Diseases; Myocarditis; Atherosclerosis | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone (Experimental): Eplerenone 50 mg twice daily along with lifestyle modification (counseling regarding diet and healthy activity) for 12 months
  Interventions: Drug: Eplerenone; Behavioral: Lifestyle Modification
- Placebo (Placebo Comparator): Placebo twice daily along with lifestyle modification (counseling regarding diet and healthy activity) for 12 months
  Interventions: Drug: Placebo; Behavioral: Lifestyle Modification

INTERVENTIONS:
Drug: Eplerenone — Eplerenone 50mg by mouth twice daily
  Arms: Eplerenone
Drug: Placebo — Placebo by mouth twice daily
  Arms: Placebo
Behavioral: Lifestyle Modification — Counseling regarding diet and healthy activity

SUMMARY:
HIV-infected individuals treated with antiretroviral medications are living longer, but have an increased risk of heart disease when compared to non-HIV-infected individuals. A hormone called aldosterone, which regulates blood pressure and sodium balance, is elevated in the HIV population in association with with increased belly fat and altered glucose metabolism. Elevations in aldosterone hormone may also be associated with abnormal blood flow, inflammation, and coronary plaque in the heart. This study is being conducted to evaluate whether therapies to reduce the actions of aldosterone may decrease the burden and progression of heart disease in the HIV population.

DETAILED DESCRIPTION:
This is a 12 month randomized, placebo controlled study enrolling HIV-infected individuals with no known history of cardiovascular disease. Eplerenone is a mineralocorticoid receptor antagonist, which can block aldosterone activation. This medication is approved by the FDA for high blood pressure and heart failure. This study aims to investigate the effect of eplerenone on other measures of cardiovascular disease in HIV. Using PET, MRI, and CT imaging technology, this study will evaluate whether eplerenone can improve coronary flow reserve and myocardial inflammation/fibrosis, in addition to atherosclerotic plaque build-up among the HIV population. The study also includes teaching on lifestyle modification to promote a healthy diet and exercise program.There are 3 overnight visits in addition to safety visits.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 40-65 years
2. Antiretroviral use (ART) >12 months and HIV viral load <100 copies/mL
3. VAT> 110cm2

Exclusion Criteria:

1. Antihypertensive use including, ACE Inhibitor, ARB, MR blockade, diuretic, potassium (K) supplementation; or BP>140/90 mmHg. Stable use (>3 months) of beta-blockers or calcium channel blockers (CCB) (except verapamil) is allowed.
2. Unstable statin use <12 months. Stable use (>12 months) is allowed.
3. Use of full dose ritonavir, nelfinavir, clarithromycin, and other strong inhibitors of CYP3A4, as well as CYP3A4 inducers.
4. Continuous oral steroid use (equivalent to prednisone > 5 mg daily) within the last 3 months.
5. Uncontrolled diabetes requiring insulin and/or HbA1c > 7.5%.
6. Creatinine (Cr) > 1.5 mg/dL or estimated GFR<60 mL/min/1.73m2.
7. K > 5.5 mEq/L.
8. Hemoglobin < 10 g/dL.
9. Known liver disease or ALT >3x ULN.
10. History of congestive heart failure, stroke, myocardial infarction, or known coronary artery disease.
11. Pregnant, actively seeking pregnancy or breastfeeding.
12. Estrogen, progestin derivative, or other sex steroid use within last 3 months. Stable physiologic testosterone replacement (> 3 months) is acceptable.
13. Current bacterial or other infections.
14. Active substance abuse.
15. Significant radiation exposure over the course of the year prior to randomization (e.g., radiation therapy, PCI, catheter ablation of arrhythmia) within 12 months of randomization.
16. Previous reaction or contraindication to iodine-containing contrast media and gadolinium.
17. Coronary artery luminal narrowing >70% on coronary CTA.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01; Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Srinivasa S, Fitch KV, Wong K, Torriani M, Mayhew C, Stanley T, Lo J, Adler GK, Grinspoon SK. RAAS Activation Is Associated With Visceral Adiposity and Insulin Resistance Among HIV-infected Patients. J Clin Endocrinol Metab. 2015 Aug;100(8):2873-82. doi: 10.1210/jc.2015-1461. Epub 2015 Jun 18. PMID 26086328
- [Derived] Walpert AR, Gupta M, Dunderdale CN, Haptu HH, Manandhar M, deFilippi CR, Burdo TH, Lee H, Kwong RY, Srinivasa S. Exploring the PREVENT HF score and myocardial function among persons with HIV. AIDS. 2025 Sep 1;39(11):1592-1597. doi: 10.1097/QAD.0000000000004252. Epub 2025 Jun 4. PMID 40478895
- [Derived] Srinivasa S, Walpert AR, Huck D, Thomas TS, Dunderdale CN, Lee H, Dicarli MF, Adler GK, Grinspoon SK. Coronary Microvascular Dysfunction Is Present Among Well-Treated Asymptomatic Persons With HIV and Similar to Those With Diabetes. Open Forum Infect Dis. 2024 Apr 26;11(5):ofae234. doi: 10.1093/ofid/ofae234. eCollection 2024 May. PMID 38813261
- [Derived] Srinivasa S, Abohashem S, Walpert AR, Dunderdale CN, Iyengar S, Shen G, Jerosch-Herold M, deFilippi CR, Robbins GK, Lee H, Kwong RY, Adler GK, Tawakol A, Grinspoon SK. Mineralocorticoid Receptor Antagonism by Eplerenone and Arterial Inflammation in HIV: The MIRABELLA HIV Study. JAMA Cardiol. 2024 Feb 1;9(2):189-194. doi: 10.1001/jamacardio.2023.4578. PMID 38090987
- [Derived] Thomas TS, Dunderdale C, Lu MT, Walpert AR, Shen G, Young MCH, Torriani M, Chu JT, Haptu HH, Manandhar M, Wurcel A, Adler GK, Grinspoon SK, Srinivasa S. Visceral Adiposity Index as a Measure of Cardiovascular Disease in Persons With Human Immunodeficiency Virus. Open Forum Infect Dis. 2023 Jul 24;10(8):ofad398. doi: 10.1093/ofid/ofad398. eCollection 2023 Aug. PMID 37559752
- [Derived] Srinivasa S, Walpert AR, Thomas TS, Huck DM, Jerosch-Herold M, Islam S, Lu MT, Burdo TH, deFilippi CR, Dunderdale CN, Feldpausch M, Iyengar S, Shen G, Baak S, Torriani M, Robbins GK, Lee H, Kwong R, DiCarli M, Adler GK, Grinspoon SK. Randomized Placebo-Controlled Trial to Evaluate Effects of Eplerenone on Myocardial Perfusion and Function Among Persons With Human Immunodeficiency Virus (HIV)-Results From the MIRACLE HIV Study. Clin Infect Dis. 2023 Oct 13;77(8):1166-1175. doi: 10.1093/cid/ciad310. PMID 37243345

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eplerenone | Placebo
Started | 20 | 20
Completed | 14 | 19
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eplerenone | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (7) | 56 (6) | 55 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 15 | 18 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 11 | 11 | 22
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Perfusion by PET
Description: Change (value at 12 months minus value at baseline) in myocardial perfusion assessed by coronary flow reserve measured via cardiac positron emission tomography. Coronary flow reserve is given by the ratio of blood flow at stress during maximal dilation of the coronary arteries to blood flow at rest.
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
unitless | 0.01 (0.64) | -0.07 (0.48)
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.72, t-test, 2 sided — P value for Change in Coronary Flow Reserve on Cardiac PET

2. Primary Outcome: Myocardial Perfusion by MRI
Description: Change (value at 12 months minus value at baseline) in myocardial perfusion assessed by myocardial blood flow measured via cardiac magnetic resonance imaging
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Mean (Standard Deviation); unit: mL/min/g
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
mL/min/g | 0.09 (0.56) | -0.53 (0.68)
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.03, t-test, 2 sided — P value for Change in Stress Myocardial Blood Flow on Cardiac MRI

3. Primary Outcome: Myocardial Inflammation
Description: Change (value at 12 months minus value at baseline) in myocardial inflammation measured by extracellular mass index (a measure of the inflammation within the heart) via cardiac magnetic resonance imaging
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: g/m^2
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
g/m^2 | 0.9 [-2.3 to 4.3] | -0.7 [-2.2 to -0.1]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.38, Kruskal-Wallis

4. Secondary Outcome: Coronary Plaque
Description: Change (value at 12 months minus value at baseline) in coronary plaque measured via coronary computed tomography angiogram assessed by coronary calcium score Scale: minimum 0 to maximum no limit, higher score indicates more plaque
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
score on a scale | 0 [0 to 6] | 5 [0 to 41]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.09, Kruskal-Wallis

5. Secondary Outcome: Markers of Vascular Dysfunction
Description: Change (value at 12 months minus value at baseline) in serum hs-cTnT
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
ng/L | 0.00 [-0.13 to 0.00] | 0.00 [0.00 to 0.74]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.03, t-test, 2 sided; Analyses performed on log transformation of data

6. Secondary Outcome: Markers of Systemic Inflammation hsIL-6
Description: Change (value at 12 months minus value at baseline) in plasma hsIL-6
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
pg/mL | -0.8 [-1.8 to 0.4] | 0.2 [-0.5 to 2.2]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.09, t-test, 2 sided — P value for Change in Plasma IL-6; Analyses performed after log transformation of data

7. Secondary Outcome: Markers of Systemic Inflammation hsCRP
Description: Change (value at 12 months minus value at baseline) in plasma hsCRP
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
ng/mL | 189 [-3841 to 718] | 591 [-261 to 2346]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.36, t-test, 2 sided — P value for Change in Plasma hsCRP; Analyses performed after log transformation of data

8. Secondary Outcome: Markers of Immune Activation MCP-1
Description: Change (value at 12 months minus value at baseline) in plasma MCP-1
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
pg/mL | 285 [49 to 365] | 292 [241 to 352]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.88, t-test, 2 sided — P value for Change in Plasma MCP-1; Analyses performed after log transformation of data

9. Secondary Outcome: Markers of Immune Activation sCD163
Description: Change (value at 12 months minus value at baseline) in plasma sCD163
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
ng/mL | -275 [-384 to -11] | -160 [-304 to 100]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.17, t-test, 2 sided — P value for Change in Plasma sCD163; Analyses performed after log transformation of data

10. Secondary Outcome: Markers of Subclinical Injury
Description: Change (value at 12 months minus value at baseline) in serum NT-proBNP
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
ng/L | 19.4 [6.6 to 41.0] | 2.8 [-25.6 to 63.5]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.28, t-test, 2 sided; Analyses performed after log transformation of data

11. Secondary Outcome: Markers of Fibrosis
Description: Change (value at 12 months minus value at baseline) in myocardial fibrosis measured by T1 (a signal intensity that measures fibrosis) via cardiac magnetic resonance imaging
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
ms | 25 [5 to 74] | 1 [-50 to 85]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.32, Kruskal-Wallis

12. Secondary Outcome: Arterial Inflammation
Description: Percentage change (value at 12 months minus value at baseline) in target to background ratio (a measure of arterial inflammation) of the index vessel measured via positron emission tomography/computed tomography
Time Frame: 12 Months
Population: Analyses performed on data available as part of a substudy.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 13 | 13
percentage change | -12.4 [-21.9 to -2.6] | 5.1 [-1.6 to 11.0]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.003, Kruskal-Wallis

13. Secondary Outcome: Markers of Arterial Inflammation
Description: Change (value at 12 months minus value at baseline) in plasma LpPLA2
Time Frame: 12 Months
Population: Analyses performed on data available as part of a substudy.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 13 | 13
ng/mL | 3.0 [-6.6 to 25.0] | 2.6 [-10.1 to 9.5]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.73, Kruskal-Wallis

14. Secondary Outcome: Assessment of Cardiac Structure by Left Ventricular Mass on Cardiac Imaging
Description: Change (value at 12 months minus value at baseline) in left ventricular mass on cardiac magnetic resonance imaging
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
g | 1 [-25 to 26] | 9 [-3 to 17]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.56, Kruskal-Wallis

15. Secondary Outcome: Assessment of Cardiac Systolic Function Via Cardiac Imaging
Description: Change (value at 12 months minus value at baseline) in global circumferential strain (GCS) on cardiac magnetic resonance imaging
Time Frame: 12 Months
Population: Analyses performed on data available
Measure: Median (Inter-Quartile Range); unit: percentage GCS
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
percentage GCS | -1.3 [-2.9 to 1.0] | 2.3 [-0.4 to 4.1]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.03, Kruskal-Wallis

16. Secondary Outcome: Assessment of Cardiac Diastolic Function Via Cardiac Imaging
Description: Change (value at 12 months minus value at baseline) in left ventricular end diastolic volume on cardiac magnetic resonance imaging
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 14 | 19
mL | -13 (28) | 10 (26)
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Test type: Superiority; p = 0.03, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Eplerenone | Placebo
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 12/20 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eplerenone (N=20) | Placebo (N=20)
Medical condition leading to death (Social circumstances) | 1 | 0 — Unrelated to study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eplerenone (N=20) | Placebo (N=20)
Dizziness (Cardiac disorders) | 4 | 0
Gastrointestinal Symptoms (Gastrointestinal disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Other Infection (Infections and infestations) | 5 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Cardiovascular Symptoms (Cardiac disorders) | 2 | 3
Injuries (Injury, poisoning and procedural complications) | 2 | 3
Other Respiratory Symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Urinary Volume Increase (Renal and urinary disorders) | 2 | 0
Underwent Non-Cardiac Elective Procedure (Surgical and medical procedures) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT02740179/Prot_SAP_000.pdf